CLINICAL TRIAL: NCT06286917
Title: Initiation of Noninvasive Ventilation in ALS Patients With Chronic Respiratory Insufficiency
Acronym: InNIVALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Heidi Rantala, Consultant, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R24001
Record Dates: First submitted 2024-02-17; First posted 2024-02-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ventilation Therapy; ALS; Chronic Respiratory Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV initiation in outpatient clinic in patients with ALS (Active Comparator): Starting the NIV at the outpatient clinic
  Interventions: Other: NIV initiation in patients with ALS
- NIV initiation in pulmonary ward in patients with ALS (Active Comparator): Starting the NIV in the pulmonary ward
  Interventions: Other: NIV initiation in patients with ALS

INTERVENTIONS:
Other: NIV initiation in patients with ALS — NIV initiation according to standard care

SUMMARY:
This research will study whether noninvasive ventilation (NIV) used to treat chronic respiratory insufficiency in patients with amyotrophic lateral sclerosis (ALS) can be initiated as successfully in the outpatient setting as in the conventional inpatient setting, and what the costs of these alternative initiation methods are.

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosed by a neurology and
* chronic respiratory insufficiency or significant respiratory muscle weakness caused by ALS

Exclusion Criteria:

* impaired cognition to give informed consent to participation
* contraindication to NIV therapy
* another severe disease with a prognosis of less than one year
* ventilation via an artificial airway, tracheostomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
NIV usage hours according to different initiation locations in patients with ALS | 5 years
  NIV daily usage hours in the 3-month control after initiation (determined over the preceding month)
Compliance with NIV according to NIV initiation setting in patients with ALS | 5 years
  Association between the initiation method and the patients' compliance with the goal of using NIV more than 4 hours per day.
Decrease in blood carbon dioxide levels in patients with ALS depending on the place of NIV initiation. | 5 years
  The effectiveness of the treatment on the reduction of blood carbon dioxide pressure

OTHER OUTCOMES:
Costs of initiation of NIV in outpatient setting compared with inpatient setting in patients with ALS | 5 years
  How much does the initiation of NIV cost in outpatient setting compared with initiation in a pulmonary ward including all the contacts with a nurse and a doctor during the following year after the initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No